CLINICAL TRIAL: NCT02590549
Title: Complete Corneal Ring (MyoRing) Implantation Combined With Corneal Collagen Crosslinking for Keratoconus
Brief Title: MyoRing Implantation With Corneal Collagen Crosslinking for Keratoconus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ufa Eye Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Myoring_CXL
Record Dates: First submitted 2015-10-25; First posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Keratoconus
Keywords: Keratoconus; riboflavin; corneal collagen crosslinking; intrasromal ring
MeSH Terms: conditions — Keratoconus | interventions — Corneal Cross-Linking

ARMS (1):
- MyoRing Implantation combined with corneal cross linking (Experimental): Surgical technique: Implantation of a MyoRing in a corneal pocket was performed by using a PocketMaker microkeratome a guided, vibrating diamond blade to create a stromal pocket 9 mm in diameter at a 300-μm depth via a 4- to 5-mm-wide corneal tunnel followed by Corneal Collagen Crosslinking (standard surface UVA irradiation (370 nm, 3 mW/cm2) using Ufalink device)
  Interventions: Procedure: Corneal Collagen Crosslinking; Device: Ufalink

INTERVENTIONS:
Procedure: Corneal Collagen Crosslinking — Sterile riboflavin solution 0.1% was then continuously injected for 3 minutes into the corneal pocket via a standard 0.3-mm cannula through the incision tunnel.
  Standard surface UVA irradiation (370 nm, 3 mW/cm2) was then applied at a 5-cm distance for 30 minutes.
  After UVA irradiation, a flexible MyoRing intracorneal implant was inserted into the corneal pocket,
Device: Ufalink — UVA irradiation with wave length 370 nm, 3 mW/cm2 is provided with UFalink, device,Russian Federation

SUMMARY:
A complete intrastromal ring, MyoRing (Dioptex, GmbH, Linz, Austria), suggested by Albert Daxer in 2007, is a relatively new technique that has been demonstrated to treat keratoconus safely and effectively.Corneal collagen crosslinking (CXL), introduced by Wollensak et al. in 2003, has become a standard treatment for progressive keratoconus to slow or possibly stop progression of disease.

The formation of the stromal pocket during MyoRing implantation offers the opportunity for simultaneous introduction of riboflavin 0.1% into the pocket followed by UVA irradiation to provide combined treatment in patients with progressive keratoconus.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* a diagnosis of keratoconus, intolerance for contact lenses or glasses
* a documented progression of disease. This progression was defined by the following changes over 1 year: an increase of the steepest K by 1.0 diopter (D) or more in manifest cylinder, or an increase of 0.5 D or more in manifest spherical equivalent (SE) refraction by repeated keratotopography ODP-scan ARK-1000 (Nidek, Japan)

Exclusion Criteria:

* minimal pachymetry of less than 380 μm,
* a history of previous ocular pathology or ocular surgery;
* pregnancy or breastfeeding;
* corneal scarring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
K max | 2 years
  Using topography measurements, decrease of maximum keratometry value over the preoperative maximum keratometry value

SECONDARY OUTCOMES:
Visual acuity as assessed by Decimal system | 2 years
  Decimal visual acuity assessed on a study later was converted to the logarithm of minimal angle of resolution (logMAR).

CONTACTS AND LOCATIONS:
Overall Officials: Mukharram Bikbov, Professor, Study Chair — Ufa Eye Research Institute

REFERENCES:
- [Background] Jadidi K, Mosavi SA, Nejat F, Naderi M, Janani L, Serahati S. Intrastromal corneal ring segment implantation (keraring 355 degrees ) in patients with central keratoconus: 6-month follow-up. J Ophthalmol. 2015;2015:916385. doi: 10.1155/2015/916385. Epub 2015 Jan 5. PMID 25685395